CLINICAL TRIAL: NCT05365529
Title: Feasibility and Efficacy of Time-Restricted Eating in Diabetes Management
Brief Title: Time-Restricted Eating for Type II Diabetes: TRE-T2D
Acronym: TRE-T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 801955
Record Dates: First submitted 2022-03-10; First posted 2022-05-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2; Time Restricted Feeding; Diabetes Type2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting | interventions — Standard of Care; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Placebo Comparator): The participants in this arm will receive the standard health and nutritional wellness guidelines and will be required to log food entries through the use of a smartphone app.
  Interventions: Behavioral: Standard of Care
- Time-Restricted Eating (Experimental): The participants in this arm will limit the number of hours they eat in day to a 8-10-hour window and will also receive the standard health and nutritional wellness guidelines. They will also be required to log food entries through the use of a smartphone app.
  Interventions: Behavioral: Time-Restricted Eating

INTERVENTIONS:
Behavioral: Time-Restricted Eating — Participants in the TRE group with continue to follow their physicians treatment plan for type II diabetes mellitus and consume all of their food within an 8-10 hour eating window.
  Other Names: Time Restricted Feeding
  Arms: Time-Restricted Eating
Behavioral: Standard of Care — Participants in the Standard of Care group will continue to follow their physician's treatment plan for type II diabetes mellitus.
  Other Names: Control group
  Arms: Standard of Care

SUMMARY:
This is a randomized clinical trial to assess the feasibility and efficacy of time-restricted eating (TRE) to improve glucose regulation and cardiovascular health of participants with type 2 diabetes mellitus (T2DM). Participants will be randomized into 2 groups: 1) standard of care (SOC), in which they will continue to follow their physician's treatment plan, or 2) SOC and TRE (8-10 hours eating window).

DETAILED DESCRIPTION:
The intervention will last for 12 weeks with a follow-up assessment at 6 months. This study will deliver the intervention, monitor participant health for safety, and promote compliance through clinic visits, virtual consultations, and an innovative combination of sensors, including continuous glucose monitors, actiwatches (to assess activity and sleep patterns), and the myCircadianClock smartphone app (to capture food, beverage, and medicine intake in real time). In-depth clinical and analytical measurements will be conducted at baseline and at the end of the intervention. We hypothesize that TRE will result in improved glucose levels (assessed via Hemoglobin A1c, the gold standard in clinical trials of T2D) and improved cardiovascular health (assessed via LDL or "bad" Cholesterol and Triglycerides). We will also be examining long-term adherence to TRE and improvements in quality of life. The proposed study will be the first adequately powered, randomized trial of TRE in patients with T2DM on background medical therapy. It is founded on a strong scientific premise and utilizes rigorous study design, state-of-the-art methods for analyzing outcomes, and an innovative approach for engaging and sustaining participation. Successful completion of this clinical trial will lay the scientific foundation and establish safety parameters for widespread implementation of TRE in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria

1. Age: 18-75 years old
2. Patients with T2DM with A1c between 6.5 and 9.0 % and on stable doses of medications who are weight-bearing and self-ambulatory.
3. Own a smartphone (Apple iOS or Android OS)
4. Baseline eating period ≥12 hours/day and sufficient logging on the mCC app.
5. Women of childbearing age will be given a pregnancy test on study enrollment and asked to use contraception throughout the study.
6. Post-menopausal and women on hormone replacement therapy will be included.
7. Estimated Glomerular Filtration Rate (EGFR) > 30mL/min/1.73m2
8. If participants are on cardiovascular medications (HMG CoA reductase inhibitors (statins), other lipid-modifying drugs, anti-hypertensives) no dose adjustments will be allowed during the study period
9. Patients on stable doses of GLP-1 receptor agonists will be included.

   Exclusion Criteria
10. Participants with Type1DM and T2DM who are taking insulin, sulfonylureas, or have an HbA1c > 9 %.
11. BMI > 50 kg/m2
12. Systolic BP greater than 160 mmHg and/or Diastolic BP greater than 110 mmHg (with or without treatment/medication)
13. LDL cholesterol greater than 200 mg/dL
14. Triglycerides greater than 500 mg/dL
15. Active tobacco or illicit drug use
16. Pregnant or breastfeeding women.
17. Currently enrolled in a weight-loss or weight-management program,
18. Currently on a special or prescribed diet for other reasons (e.g., Celiac disease),
19. The recent initiation, within the 3 preceding months prior to study enrollment, of medications designed for weight loss or with recognized appetite-suppressant effects (e.g. GLP-1 receptor agonists). Patients that are stable on such medications for at least 3 months can still be enrolled.
20. History of eating disorder(s).
21. History of surgical intervention for weight management (e) active eating disorder.
22. Chronic kidney disease with an eGFR calculated based on the Modification of Diet in Renal Disease (MDRD) equation < 30mL/min/1.73m2
23. Treatment for active inflammatory and/or rheumatologic disease and cancer.
24. A major adverse cardiovascular event within the past 6 months such as acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack (TIA).
25. History of Uncontrolled arrhythmia (i.e., rate-controlled atrial fibrillation/atrial flutter are not exclusion criteria)
26. Liver cirrhosis and/or significant alterations in liver function
27. History of (a) thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e., hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion),
28. Known inflammatory and/or rheumatologic disease.
29. Shift workers with variable (e.g., nocturnal) hours.
30. Caregivers for dependents requiring frequent nocturnal care/sleep interruptions.
31. More than one trip planned to travel to a time zone with greater than a 3-hour difference during study period.
32. History of major adverse cardiovascular events within the past 1 year (acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack (TIA)).
33. History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e., hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion).
34. History of adrenal disease.
35. History of malignancy undergoing active treatment, except non-melanoma skin cancer.
36. Known history of type I diabetes.
37. History of stage 4 or 5 chronic kidney disease or requiring dialysis.
38. History of HIV/AIDS.
39. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Glycemic regulation assessed by HbA1c | Baseline and 3 months
  Change in blood glucose assessed via hemoglobin A1c.

SECONDARY OUTCOMES:
Glycemic regulation assessed by Continuous Glucose Monitor (CGM) | Baseline and 3 months
  Change in glycemic regulation as assessed by CGM from interstitial glucose with outcomes including time in range, glycemic variability, and mean glucose.
Fasting plasma glucose (mg/dL) | Baseline and 3 months
  Change in glycemic regulation as assessed fasting plasma glucose (mg/dL).
Fasting plasma insulin (mIU/L) | Baseline and 3 months
  Change in glycemic regulation as assessed changes in fasting plasma insulin (mIU/L).
HOMA-IR | Baseline and 3 months
  Change in glycemic regulation as assessed by HOMA-IR.
LDL Particle Number (nmol/L) | Baseline and 3 months
  Changes in atherogenic lipids assessed via LDL Particle Number (nmol/L) via NMR Lipoproteinprofile.
Non-HDL Cholesterol (mg/dL) | Baseline and 3 months
  Changes in atherogenic lipids assessed via Non-HDL Cholesterol (mg/dL).
Triglycerides (mg/dL) | Baseline and 3 months
  Changes in atherogenic lipids assessed via Triglycerides (mg/dL).
Apolipoprotein B (ApoB) | Baseline and 3 months
  Changes in atherogenic lipids assessed via ApoB (mg/dL).
Quality of life Assessment via Short Form-36 Questionnaire (SF-36) | Baseline and 3 months
  Changes in quality of life as assessed by the SF-36 questionnaire.

OTHER OUTCOMES:
Safety of 8-10 hour TRE in patients with type II diabetes mellitus on stable medication assessed by daily fasting glucose and ketone measurements (finger pricks). | Baseline through 3 months
  Any hypoglycemic events reported from daily finger pricks will be reported
Long term TRE adherence | 3-month to 6-month follow-up
  Ability to self-sustain TRE assessed via logging on the mCC app 2 weeks/month. [Timeframe: 3-month to 6-month follow-up]

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

REFERENCES:
- [Derived] Taub PR, Panda S. Time for better time-restricted eating trials to lessen the burden of metabolic diseases. Cell Rep Med. 2022 Jun 21;3(6):100665. doi: 10.1016/j.xcrm.2022.100665. PMID 35732151